CLINICAL TRIAL: NCT01084824
Title: A Randomized Clinical Trial Examining the Efficacy of Treatment of Cutaneous Verruca Vulgaris in Adult Patients With Combined Liquid Nitrogen Cryotherapy and Topically Applied Cantharidin
Brief Title: A Trial Examining the Treatment of Common Warts With Combination Liquid Nitrogen (LN2) and Cantharidin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Idaho Dermatology (Other)
Responsible Party: Richard Flygare, Ph.D.; Stephen Craig, M.D., North Idaho Dermatology, TUI University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NID-001
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Last update posted 2010-03-11 (Estimated); Status verified 2010-03

CONDITIONS: Verruca Vulgaris
Keywords: Warts; Verruca vulgaris; Liquid Nitrogen; Cantharidin; combination treatment
MeSH Terms: conditions — Warts | interventions — Cantharidin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Liquid nitrogen and canthardin (Active Comparator): Liquid nitrogen applied to wart(s), then cantharidin 1% topical applied afterwards.
  Interventions: Drug: Liquid nitrogen and cantharidin
- Liquid nitrogen and placebo (Placebo Comparator): Liquid nitrogen applied to wart(s) then placebo vehicle afterwards.
  Interventions: Drug: Liquid nitrogen and topical placebo

INTERVENTIONS:
Drug: Liquid nitrogen and cantharidin — Liquid nitrogen applied to wart(s), then cantharidin 1% topical applied afterward.
  Arms: Liquid nitrogen and canthardin
Drug: Liquid nitrogen and topical placebo — Liquid nitrogen applied to wart(s), then placebo vehicle applied thereafter.
  Arms: Liquid nitrogen and placebo

SUMMARY:
The purpose of the study was to see if liquid nitrogen, a commonly used treatment for warts, is more effective if it is used alone, or if it is more effective if combined with cantharidin, a topical treatment also commonly used for warts (verruca vulgaris).

ELIGIBILITY:
Inclusion Criteria:

1. common warts on non-genital, non-facial skin
2. otherwise healthy
3. between 18-65 and able to give informed consent
4. capable of tolerating treatment

Exclusion Criteria:

1. Ill-health
2. Poor tolerance or sensitivity to treatments in study
3. <18 years old; >65 years old
4. verruca plana or condyloma acuminata
5. immunosuppression or immune dysfunction
6. significant peripheral vascular disease
7. significant sensitivity to cold
8. epidermodysplasia verruciformis
9. mosaiform warts or periungual warts

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-06; Primary Completion 2008-06 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Percentage of common warts cleared | 12 weeks
  Percentage of treated warts cleared with treatment, as measured with dermatoscopic examination, after 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Flygare, PhD, Principal Investigator — TUI University; North Idaho Dermatology
Locations (1):
- North Idaho Dermatology, Coeur d'Alene, Idaho, United States

REFERENCES:
- [Background] Berth-Jones J, Bourke J, Eglitis H, Harper C, Kirk P, Pavord S, Rajapakse R, Weston P, Wiggins T, Hutchinson PE. Value of a second freeze-thaw cycle in cryotherapy of common warts. Br J Dermatol. 1994 Dec;131(6):883-6. doi: 10.1111/j.1365-2133.1994.tb08594.x. PMID 7857844
- [Background] Guidelines of care for cryosurgery. American Academy of Dermatology Committee on Guidelines of Care. J Am Acad Dermatol. 1994 Oct;31(4):648-53. No abstract available. PMID 8089292
- [Background] Moed L, Shwayder TA, Chang MW. Cantharidin revisited: a blistering defense of an ancient medicine. Arch Dermatol. 2001 Oct;137(10):1357-60. doi: 10.1001/archderm.137.10.1357. PMID 11594862